CLINICAL TRIAL: NCT03878589
Title: Mechanisms Underlying Oxytocin's Analgesia in Older Adults
Brief Title: Understanding Cognition, Oxytocin & Pain in Elders
Acronym: UCOPE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB201801467-N; R01AG059809 (NIH); OCR18586 (Other: UF OnCore)
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: This trial will be a double-blinded, randomized crossover group design that will randomize older adults with symptomatic knee Osteoarthritis pain to four weeks of intranasal self-administration of either oxytocin (OT) or placebo (P) (48 IUs daily) followed by a four-week washout period and a second four weeks of intervention (either OT or P).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin Crossover Placebo Group (Active Comparator): During Phase 1 of the intervention, participants will self-administer via intranasal spray 24 International Units of oxytocin (OT) twice a day at home, at 8-9 in the morning and again at 5-6 in the afternoon. After a four-week washout period, Phase 2 will consist of a second four weeks of intervention, this time intranasal spray 24 International Units of placebo (P) twice a day will be self-administered.
  Interventions: Drug: Oxytocin (OT); Drug: Placebo (P)
- Placebo Crossover Oxytocin Group (Active Comparator): During Phase 1 of the intervention, participants will self-administer via intranasal spray 24 International Units of placebo (P) twice a day at home, at 8-9 in the morning and again at 5-6 in the afternoon. After a four-week washout period, Phase 2 will consist of a second four weeks of intervention, this time intranasal spray 24 International Units of oxytocin (OT) twice a day will be self-administered.
  Interventions: Drug: Oxytocin (OT); Drug: Placebo (P)

INTERVENTIONS:
Drug: Oxytocin (OT) — During the 4 week intervention, participants will self-administer twice daily 24 International Units intranasal oxytocin (OT) and will be contacted once a week for assessment of adverse effects and for download of the smartwatch data. During the last week of the intervention period, three assessment sessions will follow that will be identical to the baseline sessions.
Drug: Placebo (P) — During the 4 week intervention, participants will self-administer twice daily 24 International Units intranasal placebo (P) and will be contacted once a week for assessment of adverse effects and for download of the smartwatch data. During the last week of the intervention period, three assessment sessions will follow that will be identical to the baseline sessions.

SUMMARY:
Osteoarthritis (OA) represents a significant cause of disability worldwide and the knee is the most commonly affected joint. Oxytocin (OT) is a mediator of endogenous analgesia in animal and human studies. This proposal will test the efficacy and safety of self-administered intranasal OT over 4-weeks in older individuals relative to placebo (P) evaluating its effects on pain and function in aging and testing potential underlying neurobiological mechanisms.

DETAILED DESCRIPTION:
Osteoarthritis represents a significant cause of disability worldwide in individuals aged 65 and older, a rapidly growing segment of our population. The knee is the most commonly affected joint with pain being the primary symptom, negatively impacting physical, cognitive, and emotional functioning. Symptomatic knee osteoarthritis has been traditionally attributed to peripheral mechanisms, but measures of joint damage only modestly account for the presence or severity of osteoarthritis-related pain. The neuropeptide oxytocin has been recognized as a mediator of endogenous analgesia in animal and human studies. However, little is known about the neurobiological mechanisms underlying oxytocin's pain-relieving properties.

This study will test the efficacy and safety of self-administered intranasal oxytocin over 4-weeks in older individuals with knee osteoarthritis. Relative to placebo, daily administration of intranasal oxytocin diminished self-reported pain, physical and emotional functioning and changes in brain metabolite concentrations. With strong support from the University of Florida and the McKnight Brain Institute, this interdisciplinary project, using a comprehensive multi-methods approach, will be the first to determine the potential benefit of oxytocin as a novel analgesic therapy for knee osteoarthritis pain in aging.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis/or back pain of at least six months duration, experience pain on more days than not, with moderate pain at baseline (i.e., > 3/6 in the Visual Descriptor Scale), and who have elevated levels of plasma Imterleukin-6 (>2.5 pg/ml) will be considered for participation.

Exclusion Criteria:

* Hypersensitivity to OT or vasopressin,
* history of hyponatremia, syndrome of inappropriate antidiuretic hormone secretion, or psychogenic polydipsia,
* on vasoconstrictors such as desmopressin, pseudoephedrine, or antidiuretic medication,
* low sodium and high osmolality levels,
* excessive smoking,
* excessive drinking,
* muscle pain as a result of systemic disease,
* significant nasal pathology,
* previous or concurrent use of narcotics delivered intranasally (e.g., cocaine),
* gastroparesis.
* individuals with heart problems (e.g., cardiomyopathy, history of myocardial infarction, arrhythmias, prolonged QT interval)
* Participants will also be excluded if they have concurrent medical or arthritic conditions that could confound symptomatic knee osteoarthritis-related outcomes or coexisting disease that could preclude successful completion of the protocol including:
* systemic rheumatic condition (e.g. rheumatoid arthritis, systemic lupus erythematosus, fibromyalgia);
* a history of clinically significant surgery to the index knee;
* uncontrolled hypertension (>150/95);
* poorly controlled diabetes (HbA1c>7%);
* neurological disease (e.g., Parkinson's, Multiple Sclerosis);
* cardiovascular or peripheral arterial disease;
* serious psychiatric disorder requiring hospitalization within the past twelve months or characterized by active suicidal ideation;
* diminished cognitive function that would interfere with completion of study procedures (i.e., Montreal Cognitive Assessment score < 25)]; and
* large pieces of metal in the body or metal in the face or neck,
* claustrophobia,
* major medical surgery in the past two months,
* history of brain surgery or any serious brain condition like aneurysm, stroke, or seizures].
* pregnant individuals will be excluded

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC (Western Ontario and McMaster Universities Osteoarthritis) Index | Baseline; Week 1; Week 2; Week 3; Week 4; Week 9; Week 10; Week 11; Week 12
  Self-reported pain and function. Summary scores of the WOMAC range from 0 (No pain or disability) to 96 (Extreme pain or disability).
Change in experimental pain modulatory capacity | Baseline; Week 1; Week 2; Week 3; Week 4; Week 9; Week 10; Week 11; Week 12
  Experimental pain outcome measure is a composite score that combines conditioned pain modulation (i.e., pain inhibition) with temporal summation (i.e., pain facilitation)

SECONDARY OUTCOMES:
Change in Frontal Cortex Brain Metabolites | Baseline; Week 1; Week 2; Week 3; Week 4; Week 9; Week 10; Week 11; Week 12
  Track levels of the frontal cortex brain chemicals (tCr, MI, Cho) through use of magnetic resonance spectroscopy (MRS).

CONTACTS AND LOCATIONS:
Overall Officials: Yenisel Cruz-Almeida, PhD, MSPH, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Department of Community Dentistry and Behavioral Science, Gainesville, Florida
  - UF Health of University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cruz-Almeida Y, Montesino-Goicolea S, Valdes-Hernandez P, Huo Z, Staud R, Ebner NC. Understanding Cognition, Oxytocin, and Pain in Elders (UCOPE): protocol for a double-blinded cross-over trial in chronic knee osteoarthritis pain. Trials. 2025 Feb 7;26(1):44. doi: 10.1186/s13063-024-08715-4. PMID 39920837

DOCUMENTS (1):
  • Informed Consent Form (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03878589/ICF_000.pdf